CLINICAL TRIAL: NCT00922662
Title: Database of Patients Undergoing Cardiac Computed Tomographic Angiography (CCTA)at William Beaumont Hospital
Brief Title: Database of Patients Undergoing Cardiac Computed Tomographic Angiography at William Beaumont Hospital (CT DATABASE)
Acronym: CTDATABASE
Status: Completed | Type: Observational
Sponsor: Kavitha Chinnaiyan (Other)
Responsible Party: Sponsor-Investigator, Kavitha Chinnaiyan, Director of Cardiovascular Imaging Education, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2009-021
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: coronary artery disease; chest pain; CCTA
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to establish an overarching database of information containing historical, demographical, clinical, and intermediate and long-term outcome data from all William Beaumont Hospital (WBH) patients undergoing Cardiac Computed Tomographic Angiography (CCTA) testing for clinical or scientific reasons.

DETAILED DESCRIPTION:
The principal goal of his project is to enable the study investigators to organize WBH research activity in the field of CCTA by concentrating data from all the patients who allow use of their data in one organized, audited and securely stored database. It will allow the ability to collect retrospective and prospective data from a number of different clinical systems and securely maintain patient medical record numbers for the reference on future projects as well as identification of patients with multiple studies and multiple follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* all retrospective patients who under went a CTA and were granted a waiver of consent
* all prospective patients CTA patients who gave informed consent.

Exclusion Criteria:

* Non CTA patients
* Patients who refused participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Both genders
  * Retrospective CCTA subjects who have undergone CCTA in the past 5 years at this institution
  * Prospective subjects who will have a CCTA at this institution (ongoing)
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2008-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To establish an overarching database of information containing historical, demographical, clinical, and intermediate and long-term outcome data from all WBH patients undergoing CCTA testing for clinical or scientific reasons. | annually for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Chinnaiyan, MD, Principal Investigator — William Beaumont Hospital-Royal Oak
Locations (1):
- Beaumont Health System - Royal Oak, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No